CLINICAL TRIAL: NCT00256412
Title: Essential Fatty Acids in Management of MDD - A Pilot Study
Brief Title: Essential Fatty Acids for Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: William Coryell, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-01 200408033
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Eicosapentaenoic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Active Comparator): Low Dose
  Interventions: Drug: Eicosapentaenoic acid (EPA) 0.7 grams/day or 1.5 grams/day
- 3 (Active Comparator): High Dose
  Interventions: Drug: Eicosapentaenoic acid (EPA) 0.7 grams/day or 1.5 grams/day

INTERVENTIONS:
Drug: Eicosapentaenoic acid (EPA) 0.7 grams/day or 1.5 grams/day — Placebo and Omega 3 capsules. All participants receive 4 capsules with either 0, 2, or 4 capsules containing omega 3.
  Arms: 2; 3
Drug: Placebo — 4 capsules of placebo each day
  Arms: 1

SUMMARY:
This is a research study to determine whether omega-3 fatty acid supplementation, when taken with the antidepressant medication escitalopram (Lexapro), helps to improve depressive symptoms in individuals who have major depressive disorder (MDD).

Omega-3 fatty acids are found in foods including walnuts, some fruits and vegetables, and coldwater fish such as herring, mackerel, sturgeon, and anchovies.

DETAILED DESCRIPTION:
Primary aims

Aim 1: To determine whether measures of essential fatty acid (EFA) membrane composition predict symptom improvement during selective serotonin reuptake inhibitor (SSRI) treatment of major depressive disorder.

Aim 2: To determine whether augmentation with the EFA eicosapentaenoic acid (EPA) is likely to benefit patients who have had an inadequate improvement following four weeks of SSRI monotherapy.

Aim 3: To determine the degree to which improvement following omega-3 supplementation in SSRI partial responders reflects changes in the erythrocyte concentrations of EPA and DHA and in the ratio of EPA to arachidonic acid (AA) erythrocyte concentrations.

Secondary Aim:

To determine whether relationships between changes in tissue EFA concentrations and changes in depressive symptoms following omega-3 supplementation are mediated by changes in cytokine activity.

Primary Hypotheses:

Hypothesis 1: After four weeks of treatment with the SSRI escitalopram Montgomery-Asberg Depression Rating Scale (MADRS) scores will correlate positively with baseline RBC concentrations of EPA and DHA and negatively with baseline erythrocyte ratios of AA to EPA.

Hypothesis 2: Among patients who continue to meet criteria for MDD after four weeks of treatment, both those randomized to .7 grams and those randomized to 1.5 grams daily of EPA supplementation will show a greater mean improvement in MADRS scores after an additional six weeks than will those assigned to placebo supplementation.

Hypothesis 3: After patients who have had inadequate antidepressant responses to SSRI treatment complete six weeks of augmentation with placebo, or with .7 grams or 1.5 grams per day of EPA, a relationships will exist between final MADRS scores and both the final RBC concentrations of DHA and EPA and the final RBC ratio of AA to EPA. These relationships will resemble those between baseline RBC concentrations and subsequent responses to escitalopram and will suggest therapeutic ranges for these concentrations.

Secondary Hypothesis:

Among patients with erythrocyte EPA concentrations less than 0.82% at the beginning of the augmentation trial, the association between subsequent changes in depressive symptoms and EPA tissue concentrations will be markedly reduced by the introduction of changes in IL-1 beta, IL-10 and PGE2 into the model.

Study Design:

Phase one is a four-week open trial and is designed to test specific response predictors. A subset of subjects who complete phase one will enter phase two, a six-week, double-blind, placebo-controlled trial designed to show whether eicosapentaenoic acid (EPA) is an effective augmentation agent in patients who have had an inadequate antidepressant response.

A pilot of thirty (30) subjects, aged 18-55 years, with current major depressive disorder who have taken not regularly taken antidepressants in the previous month. Cognitively impaired subjects will not be included.

This is a pilot study designed to demonstrate the feasibility for an NIMH application. It is not currently powered to statistically test the listed hypotheses.

Study outcomes/endpoints:

The primary outcomes for both phases will be the final MADRS score.

Study Procedures:

Subjects will be recruited through advertisement and through the University of Iowa Hospitals and Clinics (UIHC) adult clinic. Advertisements will also be placed in the newspapers of cities within a 100-mile radius of UIHC.

Screening procedures:

The study's research associate will screen calls, contact respondents, and administer the screening to determine eligibility. Those who appear to satisfy entry criteria will be given appointments to meet with the PI and Co-PI. If the in-person evaluation confirms the subject's eligibility, he or she will be given a consent form and be invited to ask any remaining questions he or she might have. The protocol could begin at that visit.

Study Intervention:

Active study agents: Escitalopram and eicosupentaenoic acid (EPA). A variety of antidepressants are available for the treatment of Major Depressive Disorder (MDD). A number of psychotherapeutic approaches also have demonstrated effectiveness. Potential subjects could receive both escitalopram and EPA without participating in the study.

Placebo study agents: Placebo capsules will match the EPA capsules.

Storage:

Drug will be locked and maintained in the medical education building. Data forms and computerized data will be stored in the University of Iowa Medical Education Building. Offices and cabinets will be locked, computer files will be password protected. The lab of Arthur Spector, M.D. will analyze the blood samples.

Administration:

In phase one, subject will be given a 4 week supply of 10 mg escitalopram (Lexapro) and instructed to take one pill a day for 4 weeks.

If eligible for phase 2 of the study, subject will continue to take 10 mg of escitalopram but will also be randomly assigned to take, in addition, either 0.7 grams or 1.5grams of the EPA or a placebo.

** If depression symptoms have improved by greater than 50% at the end of week 4, subject will be given a 1 month supply of escitalopram and will be assisted in obtaining psychiatric care in their area.

If depression symptoms have not improved by greater than 50% at the end of week 4 subject will be invited to participate in Phase 2 of the study.

The protocol will begin with the administration of a structured diagnostic interview, the Structured Clinical Interview for DSM IV Diagnosis (SCID), and two depression rating scales, the Montgomery Asburg Depression Rating Scale (MADRS) and the Hamilton Rating Scale (HRS). Two tubes of blood will be drawn, one for erythrocyte EFA concentration determination and the other for quantification of inflammatory markers (c-reactive protein). Subjects will then be supplied with a one-month supply of escitalopram (Lexapro) with instructions to take one 10mg capsule each morning. Return visits at two weeks and four weeks will be scheduled and subjects will be instructed to return with any remaining medication.

Subjects will be contacted at weekly intervals. During a brief telephone conversation he or she will ask whether the subject has any questions or has experienced any troublesome side effects.

Those who meet the criteria for inadequate escitalopram response described above will be invited to participate in a six-week trial of supplemental omega-3. Subjects will continue taking escitalopram at the previous dose of 10mg daily but will be randomly assigned to take, in addition, either 0.7 grams or 1.5 grams of the eicosapentaenoic acid (EPA) or a placebo.

Visits for phase 2 will be scheduled at weeks 6, 8, and 10. At week 4 and 10 blood samples for erythrocyte EFA concentrations and cytokine determinations will be drawn. MADRS will be rated on these visits.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV criteria for nonpsychotic MDD
2. Not currently on antidepressants OR not responding to a stable dose of antidepressants

Exclusion Criteria:

1. DSM-IV for substance abuse in past month or dependence past year.
2. Allergy to fish
3. Bleeding disorder or taking warfarin
4. Omega-3 supplements for more than three consecutive days in the preceding month
5. Pregnant
6. Taking medications (i.e. glucocorticoids) known to produce affective symptoms
7. History of non-response to escitalopram
8. DSM-IV for an eating disorder in the preceding year.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) scores | 4 - 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William H Coryell, M.D., Principal Investigator — University of Iowa; Jess G Fiedorowicz, M.D., Study Director — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Appleton KM, Voyias PD, Sallis HM, Dawson S, Ness AR, Churchill R, Perry R. Omega-3 fatty acids for depression in adults. Cochrane Database Syst Rev. 2021 Nov 24;11(11):CD004692. doi: 10.1002/14651858.CD004692.pub5. PMID 34817851